CLINICAL TRIAL: NCT01722929
Title: A Pilot Study of Skin and Muscle Parameters Using a Multifunctional Skin Sensor
Brief Title: Study of Skin and Muscle Parameters Using a Skin Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology- Head and Neck Surgery and Surgery-Organ Transplantation, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU69718
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Skin Wounds

STUDY DESIGN:
Intervention Model Description: Participants had the skin sensor measure temperature both near a surgery site and also near a non-surgery site. There is one intervention (skin sensor) and the participants were assigned to both arms "surgery side" and "non-surgery side" in parallel.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Skin sensor on surgery side (Experimental): Skin sensor will be placed on the side that had surgery. This is split-body, interventional, parallel-design study. All participants will have the skin sensor measured twice on their bodies: on the side with surgery and a contralateral, control site of the body.
  Interventions: Device: Skin sensor
- Skin sensor on non-surgery side (Active Comparator): Skin sensor will be placed on the contralateral side from surgery site.This is split-body, interventional, parallel-design study. All participants will have the skin sensor measured twice on their bodies: on the side with surgery and a contralateral, control site of the body.
  Interventions: Device: Skin sensor

INTERVENTIONS:
Device: Skin sensor

SUMMARY:
The aim of this study is to assess the role of skin sensors in obtaining reliable and accurate serial measurements of skin parameters in the context of cutaneous skin wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females age 18 and over
* Recent (post-operative day 0-90) skin surgery of the trunk,extremities, head or neck for minor skin problems resulting in sutured wounds or open granulating wounds.
* Otherwise good general health as assessed by the investigator
* The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.

Exclusion Criteria:

* Under 18 years of age
* Pregnancy or Lactation
* Subjects who are unable to understand the protocol or to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-06-04 (Actual); Primary Completion 2013-09-16 (Actual); Study Completion 2013-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgery Side and Non-surgery Side: This is a split-body, parallel-designed study. All study participants had the skin sensor (the same intervention) placed near the site of their surgery wound, and also on a site without any surgery wound.
  Since this is split-body design with one intervention, participant flow will be limited to all study participants as one group to not double-count the number of participants.
Period: Overall Study
Arm/Group | Surgery Side and Non-surgery Side
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Surgery Side and Non-surgery Side: All study participants had the skin sensor placed near the site of their surgery wound, and also on a site without any surgery wound.
Arm/Group | Surgery Side and Non-surgery Side
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.75 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Measure Temperature at 3 Time Points
Time Frame: Baseline, 48 hours from baseline, and 2 weeks from baseline
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Groups:
- Skin Sensor on Surgery Side: Skin sensor will be placed on the side that had surgery.
  Sensor on surgery side.
  This is a split-body study. All participants will have the skin senor on both the surgery side and a non-surgery side.
- Skin Sensor on Non-surgery Side: Skin sensor will be placed on the contralateral side from surgery site.
  Sensor on non-surgery side
  This is a split-body study. All participants will have the skin senor on both the surgery side and a non-surgery side.
Arm/Group | Skin Sensor on Surgery Side | Skin Sensor on Non-surgery Side
Number analyzed (Participants) | 4 | 4
Degrees Celsius
  Baseline | 29.89 (0.09) | 31.13 (0.17)
  48 hrs from Baseline | 31.87 (0.35) | 32.02 (0.15)
  2 Weeks from Baseline | 33.01 (0.03) | 33.45 (0.13)
Statistical Analysis 1: Comparison: Skin Sensor on Surgery Side vs Skin Sensor on Non-surgery Side; A mixed ANOVA was performed with the arms as a between factor and the three times as the within factor; Test type: Other; p < 0.0001, Mixed Models Analysis — p-value is for the main effect for the Treatment, Time, and Treatment*Time interaction

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Surgery Side and Non-surgery Side: The skin sensor intervention was placed on both a surgery site and a non-surgery site in the same participant. This reflects all participants that received the intervention. The Arms/Groups "Surgery Side" and "Non-surgery Side" are combined because they both received the same intervention (skin sensor).
Arm/Group | Surgery Side and Non-surgery Side
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes